CLINICAL TRIAL: NCT03677687
Title: Adapting a Mindfulness-based Programme to Facilitate Physical Activity Uptake in Underactive Participants: A Feasibility Study
Brief Title: Mindfulness for Physical Activity Research Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Kat Schneider, Principal Investigator, Liverpool John Moores University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MfPA
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Physical Activity
Keywords: Mindfulness
MeSH Terms: conditions — Motor Activity | interventions — Mindfulness; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness for Physical Activity (Experimental): A 6-week mindfulness programme (2 hours per week) aimed at increasing physical activity in underactive participants.
  Interventions: Behavioral: Mindfulness for Physical Activity

INTERVENTIONS:
Behavioral: Mindfulness for Physical Activity — The Mindfulness for Physical Activity (MfPA) programme aims to change participants' relationship with physical activity by targeting psychological factors related to physical activity uptake and maintenance.

SUMMARY:
This study aims to evaluate the feasibility and preliminary effectiveness of a Mindfulness for Physical Activity programme on physical activity outcomes in underactive participants.

DETAILED DESCRIPTION:
In recent years, mindfulness-based approaches have increasingly been used in mental and physical health interventions. There appears to be some consensus about the benefits of standard mindfulness courses, such as Mindfulness-Based Stress Reduction and Mindfulness-Based Cognitive Therapy on stress, anxiety and depression, and other health conditions. In terms of physical activity, however, evidence for the use of mindfulness training to promote and improve physical activity is scarce and shows conflicting results. Evidence suggests that mindfulness training may enhance psychological factors related to exercise, such as intrinsic motivation to engage in physical activity, tolerance of physical activity-related discomfort, and physical activity self-regulation, which could potentially enhance physical activity maintenance in the long run.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 19-64 years old
* Would like to do more physical activity, but find it boring, uncomfortable, or not enjoyable
* Available and willing to attend all sessions and complete all research measures

Exclusion Criteria:

* Physical disability, cardiovascular condition, or any other illnesses or injuries that would prevent from doing physical activity
* Currently engaging in regular physical activity
* Currently taking medication and/or undergoing therapy for a mental health condition
* Have previously completed a mindfulness course
* Currently engaged in a regular meditation practice
* Away or unavailable on Mondays between 17:30 to 19:30pm for 6 weeks starting 1st October and for other assessment dates up to 17th December 2018

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility and acceptability | Up to 14 weeks
  Assessed using qualitative data gained through a focus group.

SECONDARY OUTCOMES:
Change in physical activity acceptance | Up to 14 weeks
  Measured using the Physical Activity Acceptance Questionnaire (PAAQ). The PAAQ is a 10-item measure, rated on a seven-point Likert scale, ranging from 1 (never true) to 7 (always true), with higher scores indicating higher tolerance for physical activity-related discomfort. Subscales include cognitive acceptance (e.g., "If I have the thought 'exercising today won't be enjoyable', it derails me from my exercise plan") and behavioural commitment (e.g., "Even if I have the desire to stop while I am exercising, I can still follow my exercise plan").
Change in self-reported physical activity | Up to 14 weeks
  Assessed using the International Physical Activity Questionnaire (IPAQ). The IPAQ is a 7-item measure, giving a result in multiples of resting metabolic rate (MET), with higher MET minute values indicating more physical activity. It assesses moderate-intensity physical activity, vigorous-intensity physical activity, walking, and sitting.
Change in objectively measured physical activity | Up to 14 weeks
  Assessed using accelerometers.
Change in physical activity motivation | Up to 14 weeks
  Measured using the Behavioural Regulation in Exercise Questionnaire (BREQ-3). The BREQ-3 is a 24-item measure, rated on a five-point Likert scale, ranging from 0 (not true for me) to 4 (very true for me), with higher scores indicating higher levels of motivation. Subscales include amotivation (e.g., "I don't see why I should have to exercise"), external motivation (e.g., "I exercise because other people say I should"), introjected motivation (e.g., "I feel guilty when I don't exercise"), identified motivation (e.g., "It's important to me to exercise regularly"), integrated motivation (e.g., "I exercise because it is consistent with my life goals"), and intrinsic motivation (e.g., "I exercise because it's fun").
Change in self-regulation | Up to 14 weeks
  Measured using the Brief Self-Control Scale (BSCS). The BSCS is a 13-item measure, rated on a five-point Likert scale, ranging from 1 (not at all like me) to 5 (very much like me), with higher scores indicating higher levels of self-control. Subscales include inhibition (e.g., "I am good at resisting temptation") and initiation (e.g., "I am able to work effectively toward long-term goals").
Change in dispositional mindfulness | Up to 14 weeks
  Measured using the Five Facet Mindfulness Questionnaire (FFMQ). The FFMQ is a 15-item measure, rated on a five-point Likert Scale, ranging from 1 (never or very rarely true) to 5 (very often or always true), with higher scores indicating higher levels of dispositional mindfulness. Subscales include acting with awareness (e.g., "When I do things, my mind wanders off and I'm easily distracted"), non-judging (e.g., "I criticize myself for having irrational or inappropriate emotions"), and non-reactivity (e.g., "I perceive my feelings and emotions without having to react to them").

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University Redmonds Building, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No